CLINICAL TRIAL: NCT02450357
Title: The Detection of Circulating Tumor Cells (CTCs) in Patients With Breast Cancer Undergoing Cryosurgery Combined With DC-CIK Treatment
Status: Completed | Type: Observational
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: Breast Cancer CTC 001
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Neoplastic Cells, Circulating
Keywords: Breast Neoplasms; Circulating Tumor Cells
MeSH Terms: conditions — Neoplastic Cells, Circulating; Breast Neoplasms | interventions — Flow Cytometry; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Control: Use Flow cytometry (FCM) and RT-PCR to test peripheral blood mononuclear cells(PBMCs) from healthy volunteer.
  Interventions: Other: Flow cytometry (FCM); Other: RT-PCR
- Cryosurgery group: Use Flow cytometry (FCM) and RT-PCR to test CTCs from patients who received cryosurgery only, 1 day before and 2 days after the cryosurgery.
  Interventions: Other: Flow cytometry (FCM); Other: RT-PCR
- DC-CIK treatment group: Use Flow cytometry (FCM) and RT-PCR to test CTCs from patients who received DC-CIK treatment only, 1 day before and 2 days after the DC-CIK treatment.
  Interventions: Other: Flow cytometry (FCM); Other: RT-PCR
- Cryosurgery with DC-CIK treatment group: Use Flow cytometry (FCM) and RT-PCR to test CTCs from patients received cryosurgery and DC-CIK treatment both, 1 day before and 2 days after the cryosurgery with DC-CIK treatment.
  Interventions: Other: Flow cytometry (FCM); Other: RT-PCR

INTERVENTIONS:
Other: Flow cytometry (FCM) — Use FCM to test PBMCs/CTCs from volunteers/patients.
Other: RT-PCR — Use RT-PCR to test PBMCs/CTCs from volunteers/patients.

SUMMARY:
Circulating tumor cells (CTCs) have the potential to provide a surrogate for'real-time biopsy' of tumor biological activity. Enumeration and molecular characterization of CTCs in breast cancer could play an important role in diagnosis, predicting the risk for tumor recurrence, and providing novel target therapy biomarkers. In view of these facts, the investigators wanted to demonstrate the value of multiparameter flow cytometry in detecting human tumor cells of breast cancer in normal peripheral blood after cryosurgery with or without dendritic cell(DC)-cytokine-induced killers(CIK) treatment, and the investigators also compared the specificity with reverse transcriptase polymerase chain reaction (RT-PCR) method.

DETAILED DESCRIPTION:
1 day before and 2 days after cryosurgery with or without DC-CIK treatment，approximately 17-mL ethylene diamine tetraacetic acid(EDTA)-blood was drawn by vein puncture from patients with breast cancer and healthy volunteers. The blood of the healthy volunteers will be used to evaluate the sensitivity and specificity and as negative control cells. To avoid contamination with skin cells, 2 mL blood will be discarded before the study samples will be taken.Briefly, the mononucleate cells will be separated from the blood over Ficoll- Paque for 20 min with 1800g at 4℃. The interface cells will be removed and washed, and the red blood cells(RBCs) will be removed using a lysis buffer followed by a repeated wash. The mononuclear cells will be counted and aliquot for RT-PCR and multiparameter flow cytometry on the basis of at least 2-3×106 cells for each methodology. The cell pellet will be resuspended in phosphate-buffered saline for multiparameter flow cytometry and in Trizol reagent for RT-PCR. Aim : Identification of CTCs may lead to better diagnosis and prognosis and could help to choose an adequate therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-75
2. Karnofsky performance status >60
3. Diagnosis of breast cancer based on histology or the current accepted radiological measures.
4. Classification tumor,nodes,metastasis-classification(TNM) stage: Ⅱ,Ⅲ,Ⅳ
5. Will receive cryosurgery and/or DC-CIK treatment
6. Life expectancy: Greater than 3 months
7. Patients' routine blood test, liver function and kidney function have no obvious abnormalities
8. Ability to understand the study protocol and a willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients with other primary tumor except lung cancer
2. History of coagulation disorders or anemia

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Ⅱ,Ⅲ,Ⅳ stage breast cancer come to Fuda Hospital for treatment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The number of Circulating Tumor Cells (CTCs) | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Central laboratory in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Wang HY, Ahn S, Kim S, Park S, Park S, Han H, Sohn JH, Kim S, Lee H. Detection of circulating tumor cells in patients with breast cancer using the quantitative RT-PCR assay for monitoring of therapy efficacy. Exp Mol Pathol. 2014 Dec;97(3):445-52. doi: 10.1016/j.yexmp.2014.09.003. Epub 2014 Sep 10. PMID 25217799